CLINICAL TRIAL: NCT02484573
Title: Evaluation of Intestinal Permeability in Cirrhotic Patients Before and After Treatment With Non-selective Beta Blocker (Propranolol)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAS-1116-14/15-1
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Liver Cirrhoses
Keywords: Cirrhosis; Variceal Bleeding; Non-selective beta blocker; Intestinal Permeability; Gene expression; Bacterial translocation
MeSH Terms: conditions — Fibrosis | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propanolol (Experimental): Patients will take the non-selective beta blocker propranolol for approximately 4 weeks starting immediately after endoscopy for esophageal variceal ligation. Patients will be initiated on a dose of 20mg by mouth every 12 hrs before titration to maximum tolerated dose. Patients will undergo testing before and after treatment for the variables listed in the outcomes section below.
  Interventions: Drug: Propanolol

INTERVENTIONS:
Drug: Propanolol
  Other Names: Inderalici

SUMMARY:
This study seeks to investigate whether non-selective beta blocker treatment decreases intestinal permeability in cirrhotic patients by altering the expression of genes encoding intercellular junction proteins.

DETAILED DESCRIPTION:
There is evidence that the non-selective beta-blocker (NSBB) propranolol reduces intestinal permeability and decreases bacterial translocation in cirrhotic patients, independent of hemodynamic effects on portal pressure. The mechanism by which this decrease in intestinal permeability and bacterial translocation occurs has not been established. Among the proposed mechanisms are: modification of splanchnic hemodynamics, increased gastrointestinal motility, and immunological properties of nonselective beta blockade. It is not known, however, if beta-blocker treatment decreases intestinal permeability by altering the expression of genes encoding intercellular junction proteins. This study seeks to investigate this question to improve understanding of the mechanism by which beta-blockers work in primary and secondary prophylaxis of variceal hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Diagnosis of cirrhosis of any etiology or severity as established by the treating physician (biopsy, biochemical, imaging)
* High risk gastroesophageal varices, that is those with medium/large varices or any size varices with red wale signs
* Scheduled appointment for endoscopic ligation as previously ordered by the treating physician
* Signed informed consent
* Ability to keep return appointments

Exclusion Criteria:

* Beta blocker treatment within 1 month prior to study period
* Antibiotic treatment during or within 1 month prior to study period
* Prebiotic or probiotic treatment during or within 1 month before study period
* Current immunosuppressive treatment
* Patients with active infectious process
* Patients with portal thrombosis
* Patients with hepatocellular carcinoma
* Patients with intestinal surgical shunts
* Patients with chronic diarrhea or documented celiac disease
* Patients with chronic renal failure (KDOQI: ≤ 3)
* Patients with allergy or absolute contraindication for the use of nonselective beta blockers (asthma, significant heart block, systolic BP <90 mm Hg, basal HR <55, refractory ascites)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Intestinal permeability | Baseline and after 4 weeks of propranolol treatment
  Evaluate and compare intestinal permeability using studies evaluating the absorption of three orally administered sugars (sucrose, mannitol and lactulose) in patients with cirrhosis before and after treatment with propranolol for 1 month.

SECONDARY OUTCOMES:
Expression of genes related to intestinal mucosal integrity | Baseline and after 4 weeks of propranolol treatment
  Evaluate and compare the expression of mRNA of the genes for zona occludens 1 (ZO1), occludin, claudin-1 and 2 in gastric and duodenal mucosal tissue of patients with cirrhosis, before and after treatment with propranolol for 1 month.
Presence of intercellular junction proteins by immunohistochemistry | Baseline and after 4 weeks of propranolol treatment
  Evaluate and compare the presence of intercellular junction proteins by immunohistochemistry in gastric and duodenal mucosa of patients with cirrhosis before and after treatment with propranolol for 1 month.
Serum inflammatory markers | Baseline and after 4 weeks of propranolol treatment
  Compare serum proinflammatory cytokines and lipopolysaccharide levels in patients with cirrhosis before and after treatment with propranolol for 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico